CLINICAL TRIAL: NCT06336005
Title: A First Human Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Target Engagement of Single Doses of NNC6022-0001 in Healthy Adults.
Brief Title: A Study to See How Safe a New Medicine (NNC6022-0001) is in Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6022-7683; U1111-1290-1002 (Other: World Health Organization (WHO)); 2023-505026-34 (Registry Identifier: European Medical Agency (EMA))
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers; Cardiometabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NNC6022-0001 (Experimental): Participants will be randomised to NNC6022-0001.
  Interventions: Drug: NNC6022-0001
- Placebo (NNC6022-0001) (Placebo Comparator): Participants will be randomised to placebo.
  Interventions: Drug: Placebo (NNC6022-0001)

INTERVENTIONS:
Drug: NNC6022-0001 — Participants will recieve single ascending dose (SAD) of NNC6022-0001. Dose is given in escalating manner for up to seven cohorts.
  Arms: NNC6022-0001
Drug: Placebo (NNC6022-0001) — Participants will recieve single ascending dose (SAD) of placebo. Placebo is given in escalating manner for up to seven cohorts
  Arms: Placebo (NNC6022-0001)

SUMMARY:
The study is testing a new study medicine, which is being tested as a potential medicine to treat cardiometabolic diseases.

The aim of this study is to see if the study medicine is safe, how it works in participants body, and what the body does to the study medicine.

Participants will either get NNC6022-0001 (the new study medicine) or placebo (a "dummy medicine" without the active ingredient). Which treatment participants get is decided by chance. The study medicine is a potential new medicine which cannot be prescribed by doctors.

The study will last for about 10 months in total.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women of non-childbearing potential.
2. Age 18-55 years (both inclusive) at the time of signing the informed consent.
3. Body mass index (BMI) between 18.5 to 29.9 kg/m^2 (both inclusive) at screening.
4. Body Weight: Greater than or equal to 50 kg at screening.
5. Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

1. Known or suspected hypersensitivity to study intervention(s) or similar products.
2. Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
3. Any of the below laboratory safety parameters at screening outside normal range, see designated reference range documents for specific values:.

   * Alanine Aminotransferase (ALT) above upper normal limit (UNL)
   * Aspartate aminotransferase (AST) above UNL
   * Total Bilirubin (BL) above UNL
   * Creatinine above UNL
   * International normalized ratio (INR) above UNL
   * Fibrinogen outside normal range of 1.6 - 4.2 gram pr. Liter (g/L)
   * C-reactive protein (CRP) above 5 milligram pr. Liter (mg/L) (males) and above 8 mg/L (females)
4. Use of prescription medicinal products or vaccines within 14 days before dosing and/or non prescription medicinal products within 7 days before dosing.

Exceptions are: Topical medications not reaching systemic circulation; less than once per week of over-the-counter paracetamol, ibuprofen and/or acetylsalicylic acid at their labelled doses for mild pain; vitamins at their labelled doses.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAE) | From time of dosing (Day 1) to end of study (Day 14)
  Number of events

SECONDARY OUTCOMES:
AUC0-t, SD; the area under the NNC6022 0001 plasma concentration-time curve from time 0 to last measurable plasma concentration after a single dose | From pre-dose (Day 1) to end of exposure (Day 7)
  Hours*micrometer (hr×µM)
AUC0-∞, SD; the area under the NNC6022 0001 plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose (Day 1) to end of exposure (Day 7)
  Hours*micrometer (hr×µM)
Cmax, SD; the maximum plasma concentration of NNC6022 0001 after a single dose | From pre-dose (Day 1) to end of exposure (Day 7)
  Micrometer (µM)
IL-1β, SD; ratio of <Timepoint> (time of the maximal plasma concentration of NNC6022 0001) to baseline | From pre-dose (Day 1) to estimated tmax (Day 1)
  Percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (Dept. 2834)., Study Director — Novo Nordisk A/S
Locations (1):
- ICON - location Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://www.novonordisk-trials.com